CLINICAL TRIAL: NCT05359263
Title: A 6-Month, Randomized, Double-Blind Study to Evaluate the Effect of Dapagliflozin on EChOcardiographic Measures of CarDiac StructurE and Function in Patients with Chronic Kidney Disease
Brief Title: Effects of Dapagliflozin on EChOcardiographic Measures of CarDiac StructurE and Function in Patients with CKD
Acronym: DECODE-CKD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tor Biering-Sørensen (Other)
Responsible Party: Sponsor-Investigator, Tor Biering-Sørensen, Research Director, MD, PhD, MPH, Herlev and Gentofte Hospital
Organization: Herlev and Gentofte Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DECODE-CKD
Record Dates: First submitted 2022-04-28; First posted 2022-05-03 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin 10 mg once daily (Experimental)
  Interventions: Drug: Dapagliflozin 10 mg
- Placebo once daily (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin 10 mg — The intervention arm consists of dapagliflozin 10 mg orally once daily
  Arms: Dapagliflozin 10 mg once daily
Drug: Placebo — The comparator arm consists of placebo orally once daily
  Arms: Placebo once daily

SUMMARY:
The purpose of this study is to investigate the effects of dapagliflozin on echocardiographic measures of cardiac structure and function in patients with chronic kidney disease.

DETAILED DESCRIPTION:
The study is a 6-month, investigator-initiated, randomized, double-blind, placebo-controlled clinical trial to evaluate the effects of dapagliflozin on echocardiographic measures of cardiac structure and function in patients with chronic kidney disease. The study population will consist of approximately 222 adults with chronic kidney disease - defined as a glomerular filtration rate (GFR) of 20-60 mL/min/1.73m2, in treatment with maximally tolerated ACEi or ARB. Patients will be randomized to either 10 mg dapagliflozin or placebo. Patients will be assessed by measurement of echocardiography, pulse wave velocity, blood samples, urine samples, quality of life, depressive symptoms, and cognitive function at baseline and after 6 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* ≥ 18 years of age
* Chronic kidney disease (CKD), defined as evidence of decreased eGFR (eGFR ≥20 and <60 mL/minute per 1.73 m2) or between eGFR ≥60 and <90 mL/minute per 1.73 m2 with urinary albumin:creatinine ratio ≥200 mg/g or protein:creatinine ratio ≥300 mg/g
* Stable treatment with clinically appropriate doses of ACEi/ARB among CKD patients with proteinuria and uptitrated to maximal recommended or tolerated dose for at least 4 weeks before randomization, if not medically contraindicated
* For patients with type 2 diabetes:

Stable antihyperglycemic treatment > 30 days before screening

* Female patients should either not be of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile, or is of childbearing potential and practicing one of the following methods of contraception throughout the study and for 30 days after study completion: Hormonal contraception (oral contraceptives, contraceptive implant, injectable birth control, contraceptive patch, or vaginal ring) or intrauterine device
* Ability to understand and read Danish

Exclusion Criteria:

* Type 1 diabetes
* For patients with type 2 diabetes:

History of diabetic ketoacidosis

* Patients undergoing dialysis
* History of organ transplant
* Treatment with SGLT2 inhibitor within 8 weeks prior to enrolment
* Known allergy or hypersensitivity to SGLT2 inhibitors or Placebo ingredients
* Myocardial infarction, unstable angina, stroke or transient ischemic attack within 12 weeks of enrolment
* Coronary revascularization (percutaneous coronary intervention or coronary artery bypass grafting) or valvular repair/replacement within 12 weeks prior to enrolment
* Any condition outside the renal and cardiovascular study area with a life expectancy of <2 years based on investigator's clinical judgement
* Hepatic impairment (aspartate transaminase or alanine transaminase >3 times the upper limit of normal [ULN] or total bilirubin >2 times the ULN at the time of enrolment)
* Known blood-borne diseases, such as Hepatitis A, B, C, D, and E, and Human immunodeficiency virus (HIV) types 1 and 2, Ebola, Lassa fever virus.
* Female patients who are pregnant, lactating, or are considering becoming pregnant during the study or for 6 months after study completion
* Participation in another clinical study with an investigational product within the last month prior to enrolment
* Inability to understand or comply with the investigational product, procedures, and/or follow-up or any conditions that may prevent the participant to complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Estimated)
Dates: Start 2022-06-08 (Actual); Primary Completion 2025-02-18 (Estimated); Study Completion 2025-02-18 (Estimated)

PRIMARY OUTCOMES:
Change in LV mass index assessed by echocardiography at 6 months | 6 months

SECONDARY OUTCOMES:
Change in LVEF assessed by echocardiography at 6 months | 6 months
Change in LA volume index assessed by echocardiography at 6 months | 6 months
Change in GLS assessed by echocardiography at 6 months | 6 months
Change in high sensitivity troponin I (hs-TNI) at 6 months | 6 months
Change in N-terminal pro B-type natriuretic peptide (NT-pro-BNP) at 6 months | 6 months
Change in estimated glomerular filtration rate (eGFR) 6 months | 6 months
Change in urinary albumin-to-creatinine ratio (UACR) at 6 months | 6 months
Change in hemoglobin at 6 months | 6 months
Change in LV mass assessed by echocardiography at 6 months | 6 months
Change in LV end-diastolic volume at 6 months | 6 months
Change in LV end-systolic volume at 6 months | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Tor Biering-Sørensen, Study Chair — Research Director
Locations (1):
- Gentofte Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Bartholdy KV, Johansen ND, Skaarup KG, Modin D, Landler N, Langhoff AF, Ottosen CI, Espersen C, Dons M, Borchsenius JIM, Davodian LW, Lassen MH, Davidovski FS, Jensen AMR, Sengelov M, Christensen J, Schou M, Feldt-Rasmussen B, Jensen J, Bressendorff I, Persson F, Rossing P, Kober L, Zannad F, Vaduganathan M, Solomon S, Haynes R, Hansen D, Biering-Sorensen T. Cardiac Effects of Dapagliflozin in People with Chronic Kidney Disease. NEJM Evid. 2025 Nov;4(11):EVIDoa2500158. doi: 10.1056/EVIDoa2500158. Epub 2025 Oct 28. PMID 41147829
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- [Derived] Bartholdy KV, Johansen ND, Landler N, Skaarup KG, Jensen J, Bressendorff I, Schou M, Christensen J, Feldt-Rasmussen B, Vaduganathan M, Solomon S, Haynes R, Persson F, Rossing P, Kober L, Zannad F, Hansen D, Biering-Sorensen T. Effects of Dapagliflozin on EChOcardiographic Measures of CarDiac StructurE and Function in Patients with Chronic Kidney Disease: The DECODE-CKD Trial. Kidney360. 2023 Feb 1;4(2):143-149. doi: 10.34067/KID.0006982022. Epub 2022 Dec 18. PMID 36649484